CLINICAL TRIAL: NCT05891106
Title: AONDA Therapeutic Indication Study I
Status: Completed | Type: Observational
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Other Study IDs: CLD265-P002
Record Dates: First submitted 2023-05-24; First posted 2023-06-06 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Bullous Keratopathy; Corneal Erosion; Entropion; Corneal Edema; Corneal Dystrophy; Corneal Ulcer; Foreign Body in Cornea; Bell Palsy; Keratoconjunctivitis; Filamentary Keratitis; Sicca Syndrome; Keratoconjunctivitis (Etiology)
MeSH Terms: conditions — Entropion; Corneal Edema; Corneal Dystrophies, Hereditary; Corneal Ulcer; Bell Palsy; Keratoconjunctivitis; Sjogren's Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- AONDA Therapeutic: Lotrafilcon A contact lenses worn therapeutically as a bandage lens as instructed by the eye care professional
  Interventions: Device: Lotrafilcon A contact lenses

INTERVENTIONS:
Device: Lotrafilcon A contact lenses — CE-marked silicone hydrogel contact lenses
  Other Names: AONDA; AIR OPTIX® NIGHT & DAY® AQUA

SUMMARY:
This study will be used to support assessment of AIR OPTIX® NIGHT & DAY® AQUA (AONDA) Soft Contact Lenses' safety and performance in accordance with updated European Union Medical Device Regulation (EU MDR) requirements.

DETAILED DESCRIPTION:
In this retrospective observational study, the subject wore AONDA as a therapeutic lens for the treatment of a corneal condition with pain in one or both eyes.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of a corneal condition with pain for which AONDA Soft Contact Lens as a therapeutic contact lens was placed on one or both eye(s) at Baseline.
* Baseline and Follow-up (up to 1 year from Baseline) charts available.
* Other protocol-defined inclusion criteria may apply.

Key Exclusion Criteria:

* Had a condition (pathological, behavioral, and/or situational) that contraindicated therapeutic contact lens wear or confounds study results during the data collection period, as determined or known by the Investigator.
* Used systemic or ocular medication that would confound study results during the data collection period, as determined or known by the Investigator.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Investigators will enroll charts following a pre-identified process.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2023-06-28 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2023-07-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in corneal pain at the Follow-up Visit | Baseline, Follow-Up Visit (up to 1 year following the Baseline Visit)
  The Investigator will review the subject's chart and document change from baseline in corneal pain at the Follow-up visit as "improved, similar, or worsened." The Baseline Visit is defined as the first visit where the AONDA therapeutic contact lens was placed on eye as part of a treatment plan for an ocular condition. The Follow-up Visit is defined as the first visit where the AONDA therapeutic contact lens was removed from the eye, or the first visit following the removal of the contact lens if, for example, the contact lens was removed between visits.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Lead, CRD Vision Care, Study Director — Alcon Research, LLC
Locations (3):
- United States (3):
  - Vision Health Institute, Orlando, Florida
  - Franklin Park Eye Center PC, Franklin Park, Illinois
  - Optometry Group, PLLC, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No